CLINICAL TRIAL: NCT07080450
Title: Post-market Clinical Follow-up Study to Collect Safety, Performance and Clinical Benefits of the ComposiTCP™ Suture Anchors Double Loaded With BroadBand Tape, Sliding
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the ComposiTCP
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-197SM
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Repairs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the ComposiTCP Suture Anchors Double Loaded with BroadBand Tape, Sliding: No specific interventions will be administered.

SUMMARY:
The study is a multicenter, retrospective and prospective, non-randomized, noncontrolled, and consecutive series post-market study. The purpose of this study is collect data confirming safety, performance and clinical benefits of the ComposiTCP Suture Anchors Double Loaded with BroadBand Tape, Sliding implants when used in rotator cuff repair.

The primary endpoint of this study is the assessment of performance by analyzing soft tissue to bone healing in the shoulder (rotator cuff). Healing will be assessed by the investigator using PROMs and clinical outcomes of the patient.

The clinical benefit will be assessed by functional outcomes measured using standard and well-established scoring systems (e.g. Oxford Shoulder Score and EQ-5D-5L) at 1 year post-operative.

The safety will be assessed by monitoring the incidence and frequency of device- and/or procedure-related adverse events.

DETAILED DESCRIPTION:
The ComposiTCP Suture Anchors Double Loaded with BroadBand Tape, Sliding implants are intended for use in rotator cuff repairs. They are intended for for the reattachment of soft tissue to bone.

Up to two sites will be involved in this study. The aim is to include a total of 43 consecutive series cases who received the device. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop and immediate post-op intervals will be available in medical notes and collected retrospectively. During follow-up visits at 1 years post-op, the patient will be asked to complete patient questionnaires. Moreover, a clinical assessment will be conducted. In addition, any complications and adverse events will also be collected during these follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject was treated with the ComposiTCP Suture Anchors Double Loaded with BroadBand Tape, Sliding for rotator cuff repair;
* At least 18 years old and skeletally mature;
* Willing and able to comply with the study procedures;
* Subject is capable of understanding the doctor's explanations, following his instructions and is able to participate in the follow-up program;
* Subject is able to read and understand the ICF and has voluntarily provided written informed consent or non-opposition.

Exclusion Criteria:

* Subject is vulnerable (is unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response);
* The subject is unwilling or unable to give consent or to comply with the follow-up program;
* Subject meets any contraindications of the appropriate Instruction for Use;
* Off-Label Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must have been treated with the ComposiTCP Suture Anchors Double Loaded with BroadBand Tape, Sliding for rotator cuff repair.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of performance by analyzing soft tissue to bone healing in the shoulder (rotator cuff) | From operation to study completion, 0-1 year
  The investigator will clinically evaluate at 1 year follow-up visit if soft tissue to bone healing has occurred by the absence of device-related revisions and re-tears that were not previously reported. The following question will be asked to the investigator: "Did soft tissue to bone healing occur"? If "yes" is answered, then the soft tissue to bone healing is successful, if "no" is answered, then the soft tissue to bone healing is considered unsuccessful.

SECONDARY OUTCOMES:
EQ-5D-5L Score | From operation to study completion, 0-1 year
  Assessment of clinical benefits by functional outcomes measured using standard scoring systems. The EQ-5D measures 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a total of 5 questions. It is accompanied by the patient's self-assessment with the VAS. Each dimension is assigned one of three discrete levels for evaluation on the day of administration: Level 1 - No problems, no disability Level 2 - Some problems, moderate disability Level 3 - A lot of problems, severe disability The final score is a five digit composite of the responses ranging between 33333 - 11111 with 243 possible combinations in between
The incidence and frequency of device and/or procedure related adverse events | From operation to study completion, 0-1 year
  Safety will be assessed by monitoring the incidence and frequency of device and/or procedure related adverse events
Oxford Shoulder Score | From surgery until study completion, 0-1 year
  The OSS is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following TSA. The OSS consists of twelve questions covering function and pain associated with the shoulder. To calculate the total score, each question is scored from 5 (worst outcome) to 0 (best outcome) and the sum of all 12 items is reported with a maximum of 60, representing the worst score possible.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (1):
- Clinique Mutualiste de Bretagne Occidentale, Quimper, France